CLINICAL TRIAL: NCT07124845
Title: Focusing on the Mind: The Effectiveness of Multimedia Cases Combined With Focused Conversation in Enhancing Nursing Students' Mental Health Literacy
Brief Title: Using Multimedia Cases Combined With Focused Conversation in Enhancing Nursing Students' Mental Health Literacy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EZRPF3Q0491
Record Dates: First submitted 2025-07-31; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Mental Health; Literacy
Keywords: mental health literacy; nursing students; multimedia
MeSH Terms: conditions — Psychological Well-Being; Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants (single group) (Experimental): Receive the 8 times of multimedia cases videos with focused conversation.
  Interventions: Other: Focusing on the mind

INTERVENTIONS:
Other: Focusing on the mind — 8 times of multimedia cases videos and focused conversation

SUMMARY:
This study aims to explore the effectiveness of the multimedia cases with focused conversation in enhancing nursing students' mental health literacy.

DETAILED DESCRIPTION:
In Taiwan, more than 50% of nursing students have mental disturbance, It is important to improve nursing students' mental health literacy. Therefore, this study aims to explore the effectiveness of the multimedia cases with focused conversation in enhancing nursing students' mental health literacy. Eight multimedia cases will be developed first, then, mixed-methods will be used in this study. Research tools include demographic questionnaire and the Mental Health Literacy Scale for Healthcare Students (MHLS-HS). Participants will fill the questionnaires before and after the intervention. After the intervention, semi-structured interview guide will be used to conduct the qualitative research.

ELIGIBILITY:
Inclusion Criteria:

* willing to participate in the study
* understand the questionnaires
* age ≥ 18 years old.

Exclusion Criteria:

* people who choose this course after the intervention begins

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
mental health literacy | MHLS-HS: Baseline (pre-intervention) and after intervention ; Interviews: after intervention.
  Using Mental Health Literacy Scale for Healthcare Students (MHLS-HS) and interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University of Science and Technology, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Undecided.